CLINICAL TRIAL: NCT00801177
Title: Phase I Study of the Fully Human Anti-Epidermal Growth Factor Receptor (EGFR) Monoclonal Antibody IMC-11F8 in Patients With Solid Tumors Who Have Failed Standard Therapy
Brief Title: Study of IMC-11F8 in Patients With Tumors Who Have Not Responded to Standard Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, ImClone LLC
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 14088; 2004-002072-42 (EudraCT Number); CP11-0401 (Other: ImClone, LLC)
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Solid Tumors
Keywords: Tumors; Antibodies, Monoclonal
MeSH Terms: conditions — Neoplasms | interventions — necitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMC-11F8 (Every week) (Experimental): Cycle of therapy administered intravenously, once a week for 6 weeks, for a total of six doses per cycle.
  Interventions: Biological: IMC-11F8; Biological: IMC-11F8 I.V.
- IMC-11F8 (Every other week) (Experimental): Cycle of therapy administered intravenously, every other week for 6 weeks, for a total of three doses per cycle.
  Interventions: Biological: IMC-11F8

INTERVENTIONS:
Biological: IMC-11F8 — Cohort 1
  100 mg I.V.
  Other Names: necitumumab
  Arms: IMC-11F8 (Every week)
Biological: IMC-11F8 — Cohort 2
  200 mg I.V.
  Other Names: necitumumab
  Arms: IMC-11F8 (Every week)
Biological: IMC-11F8 — Cohort 3
  400 mg I.V.
  Other Names: necitumumab
  Arms: IMC-11F8 (Every week)
Biological: IMC-11F8 I.V. — Cohort 4
  600 mg I.V.
  Other Names: necitumumab
  Arms: IMC-11F8 (Every week)
Biological: IMC-11F8 — Cohort 5
  800 mg I.V.
  Other Names: necitumumab
  Arms: IMC-11F8 (Every week)
Biological: IMC-11F8 — Cohort 6
  1000 mg I.V.
  Other Names: necitumumab
  Arms: IMC-11F8 (Every week)
Biological: IMC-11F8 — Cohort 1
  100 mg I.V.
  Other Names: necitumumab
  Arms: IMC-11F8 (Every other week)
Biological: IMC-11F8 — Cohort 2
  200 mg I.V.
  Other Names: necitumumab
  Arms: IMC-11F8 (Every other week)
Biological: IMC-11F8 — Cohort 3
  400 mg I.V.
  Other Names: necitumumab
  Arms: IMC-11F8 (Every other week)
Biological: IMC-11F8 — Cohort 4
  600 mg I.V.
  Other Names: necitumumab
  Arms: IMC-11F8 (Every other week)
Biological: IMC-11F8 — Cohort 5
  800 mg I.V.
  Other Names: necitumumab
  Arms: IMC-11F8 (Every other week)
Biological: IMC-11F8 — Cohort 6
  1000 mg I.V.
  Other Names: necitumumab
  Arms: IMC-11F8 (Every other week)

SUMMARY:
The purpose of this study is to determine if IMC-11F8 is safe for patients, and also to determine the best dose of IMC-11F8 to give to patients.

DETAILED DESCRIPTION:
The purpose of this study is to establish the safety profile and the maximum tolerated dose (MTD) of the fully human anti-EGFR monoclonal antibody IMC-11F8 in patients with solid tumors who have filed standard therapy or for whom no standard therapy is available.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed, EGFR-detectable or EGFR-undetectable, unidimensionally-measurable and/or evaluable solid tumors who failed standard therapy or for whom no standard therapy is available. Patients who do not have tissue available for EGFR testing will undergo a biopsy of an accessible tumor.
* ECOG performance status score of ≤ 2 at study entry.
* Able to provide written informed consent.
* White blood cell (WBC) count ≥ 3 x 109/L; an absolute neutrophil count ≥ 1.5 x 109/L; a hemoglobin level > 90 g/L; and a platelet count ≥ 100 x 109/L.
* Adequate hepatic function as defined by:

  * an alkaline phosphatase level ≤ 5.0 x the ULN
  * a bilirubin level ≤ 1.5 x the ULN
  * aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤ 2.5 x the ULN or ≤ 5 x the ULN for patients with liver metastases
* Adequate renal function as defined by a serum creatinine level within normal limits.
* Use of effective contraception if procreative potential exists.
* Life expectancy of approximately 3 months in the opinion the opinion of the investigator.

Exclusion Criteria:

* Chemotherapy, radiation, and/or hormonal therapy (except palliative radiation therapy for disease-related pain and chronic hormonal therapy for prostate carcinoma) within 4 weeks of study entry.
* Concurrent unstable or uncontrolled medical disease (e.g., active uncontrolled systemic infection, poorly controlled hypertension or history of poor compliance with an anti-hypertensive regimen, unstable angina, congestive heart failure, uncontrolled diabetes) or other chronic disease, which, in the opinion of the investigator, could compromise the patient or the study.
* Newly-diagnosed or symptomatic brain metastases (patients with a history of brain metastases must have received definitive surgery or radiotherapy, be clinically stable, and not taking steroids; anticonvulsants are allowed).
* Any concurrent malignancy other than basal cell carcinoma or carcinoma in situ of the cervix. Patients with a previous malignancy but without evidence of disease for ≥ 3 years will be allowed to enter the trial.
* Any condition that prevents the patient from providing informed consent.
* Pregnancy (confirmed by serum beta human chorionic gonadotropin [ßHCG]) or breast-feeding.
* Any investigational agent(s) or device(s) within 4 weeks of study entry.
* Prior treatment with cetuximab, or any other epidermal growth factor receptor inhibitors, including tyrosine kinase inhibitors, such as gefitinib or erlotinib. Prior treatment with other monoclonal antibodies targeting receptors other than the EGFR is permitted ≥ 4 weeks prior to study entry.
* Any prior therapy that targeted the EGFR or EGFR pathway.
* Known history of human immunodeficiency virus.
* Employees of the investigator or study center with direct involvement in this study or other studies under the direction of the investigator or study center, as well as family members of the employees.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Approximately 24 Months
Maximum Tolerated Dose of IMC-11F8 | Approximately 24 Months

SECONDARY OUTCOMES:
Area under the Time Concentration Curve (AUC) | Approximately 24 Months
Maximum concentration (Cmax) | Approximately 24 Months
Half-life (t 1/2) | Approximately 24 Months
Serum Anti-IMC-11F8 Antibody Assessment | Approximately 24 Months
Change from baseline in Antitumor Activity | Approximately 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Chair — Eli Lilly and Company
Locations (2):
- Netherlands (2):
  - ImClone Investigational Site, Amsterdam
  - ImClone Investigational Site, Utrecht

REFERENCES:
- [Result] Kuenen B, Witteveen E, Ruijter R, Ervin-Haynes A, Tjin-A-ton M, Fox F, et al. A phase I study of IMC-11F8, a fully human anti-epidermal growth factor receptor (EGFR) IgG1 monoclonal antibody in patients with solid tumors. Interim results. [abstract 3024 and poster presentation]. American Society of Clinical Oncology Annual Meeting. 2006 June 2-6; Atlanta, GA.
- [Result] Kuenen B, Witteveen PO, Ruijter R, Tjin-A-Ton M, Youssoufian H, Rowinsky E, et al. A phase I study of IMC-11F8, a recombinant human anti-epidermal growth factor receptor IgG1 monoclonal antibody in patients with solid tumors. [abstract B52 and poster presentaton] International Conference on Molecular Targets and Cancer Therapeutics 2007 Oct 22-26; San Francisco, CA.